CLINICAL TRIAL: NCT02286063
Title: Randomized, Controlled Crossover Trial to Evaluate the Effects of Ambulatory Oxygen on Health Status in Patients With Fibrotic Lung Disease (FLD).
Brief Title: Ambulatory Oxygen in Fibrotic Lung Disease (FLD) (AmbOx)
Acronym: AmbOx
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2013OE005B; 2013-004355-20 (EudraCT Number)
Record Dates: First submitted 2014-10-08; First posted 2014-11-07 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Lung; Disease, Fibroid (Chronic)
MeSH Terms: conditions — Disease; Leiomyoma; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ambulatory oxygen cylinders (Active Comparator): Subjects randomised to have the intervention of portable oxygen for the first two weeks. Only patients with stable symptoms at the end of the 'run in' period and reproducible 6-minute walk distance on the 6MWT during the baseline visit, as a marker of clinical stability of the disease will be randomized. They will be a portable oxygen cylinder during 2 weeks when they realize activities.
  Interventions: Drug: Ambulatory Oxygen
- no oxygen cylinders (No Intervention): Subjects randomised to be on air for the first two weeks of the treatment period.

INTERVENTIONS:
Drug: Ambulatory Oxygen — The IMP investigated in this study is medical oxygen (PL 15929/005), manufactured by Air Liquide Ltd. UK. Oxygen is a colourless, odourless gas with molecular weight 32, a boiling point of 183.1°C (at 1 bar) and a density of 1.355 kg/m3 (at 15°C and 1013mb).
  Oxygen is present in the atmosphere at 21% and is an absolute necessity for life. Each of the four oxygen companies across the UK provide a light and a standard weight oxygen cylinder. Ambulatory Oxygen will be given to the Oxygen arm.
  Other Names: portable oxygen cylinders, light weight oxygen cylinders
  Arms: ambulatory oxygen cylinders

SUMMARY:
The main aim of this project is to establish whether ambulatory oxygen in patients with fibrotic ILD whose oxygen saturation falls ≤ 88% on a 6MWT, leads to a significant improvement in health status. The core of the project will be a four week randomised, crossover controlled trial of ambulatory oxygen used during daily activities. The optimal Oxygen flow rate is determined by titration at screening visit and administered during activity for a two-week period, compared to two weeks off oxygen.

DETAILED DESCRIPTION:
The planned non-commercial study is a randomised, controlled crossover trial of ambulatory oxygen against no ambulatory oxygen over a four week period (two weeks on ambulatory oxygen and two weeks on air, with no portable devices), to evaluate the effects of ambulatory oxygen on health status in patients with ILD. A short crossover study in this context has many advantages, since ambulatory oxygen has immediate effect, with no wash-out period needed after use. The primary outcome of the study will be the change in health status, as measured by the K-BILD questionnaire (Thorax 2012 67: 804-810).

At the start of the trial, the effects of ambulatory oxygen on 6 Minute Walk Test (6MWT) parameters will be evaluated on oxygen and on air-filled canisters, with the patient blind to the contents of the canister, to assess whether oxygen-induced improvements in 6MWT parameters can predict its effectiveness in day to day life. The 6MWT is a well established and highly reproducible test validated in ILD patients, with significant prognostic implications.

The study design does not include a placebo arm because:

1. The intervention is a combination of possible benefits from oxygen and the disadvantage of canister weight. These cannot be separated. Placebo control is impossible because there is no means of providing placebo weight. Attempts to control solely for oxygen use without taking canister weight into account are clinically meaningless. In a recent COPD, chronic obstructive pulmonary disease study, cylinder weight was reported as a barrier to use by 93% of study participants.
2. A positive result against an air-filled canister arm would be clinically uninterpretable. This is a study design in which the 'placebo' would be actively harmful to study participants. Carriage of an air-filled cylinder would be expected to lead to earlier desaturation and reduced exercise tolerance. Such a design would not inform the real life comparison between oxygen plus cylinder and no intervention.
3. All this aside, blinding is legally impossible (UK health and safety regulations require that oxygen cylinders for home use must be clearly labelled).

It should also be stressed that objective measures of change are evaluated as secondary end-points: the investigators expect to explore correlations between these variables and the primary end-point to exclude the possibility that an observed treatment benefit on the primary end-point might be confounded by a placebo effect.

A more in depth qualitative assessment of the impact of ambulatory oxygen will be undertaken via a semi-structured interview, in a subset of 20 patients, to investigate patients' and their carers' personal perspective on how the ambulatory oxygen has affected their day to day life. The interview will be conducted within 2 weeks of the end of treatment visit. Patients from the Royal Brompton Hospital site will be approached by the researcher at the end of treatment visit and asked if they will participate in the qualitative assessment. If the patient agrees a date will be agreed for the patient to be interviewed at a venue convenient to them (usually the patient's home).

During the interviews a semi-structured topic guide will address practical barriers to optimal oxygen usage, practical, social and psychological difficulties encountered, concerned about dependency, and views on the information required prior to ambulatory oxygen prescription. The interviews will also explore patients' (and carers') experience of participating in the trial. Notes will be written after each interview to aid reflective analytical processes. Individual feed back on how the system and the service could be improved will assess how the needs of patients and their future involvement can be incorporated into the design of more patients and their future involvement can be incorporated into the design of more patients centred devices.

Qualitative interview analysis: Interviews will be transcribed verbatim. Interview transcripts will be analysed thematically using a framework approach. Atlas/ti computer software (http://atlasti.com) will be used to manage and index the data prior to charting, mapping and interpretation.

ELIGIBILITY:
Inclusion Criteria:

* IPF or another fibrotic ILD (including fibrotic NSIP, fibrotic organising pneumoni, and fibrotic hypersensitivity pneumonitis)
* patients aged 18 - 99 yrs
* Desaturation ≤ 88% on a 6MWT on room air
* Stable respiratory symptoms in the 4 weeks preceding the trial including the run in period

Exclusion Criteria:

* Patients meeting criteria for long term oxygen therapy, including hypercapnic patients
* Patients expected to change treatment during the course of the study
* Significant locomotor or communication difficulties and/or severe co-morbidities
* Patients with sarcoidosis or connective tissue disease affecting the musculoskeletal system
* Current smokers
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-08; Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
change in K-BILD The King's Brief Interstitial Lung Disease Questionnaire health status score | February 2017 (up to 3 years)
  The mean change vs baseline in the K-BILD health status score on and off ambulatory oxygen will be compared by using either a paired t-test or Wilcoxon signed rank test, as appropriate to the distribution of the data. To allow assessment of the effect of baseline values on treatment and any other potential confounders, regression with robust variances or linear mixed models will be used. STATA software will be used for statistical analysis.

SECONDARY OUTCOMES:
Dyspnoea scores | 2 weeks
  assessed by the San Diego shortness of breath questionnaire.
Global assessment of change in walking ability and exertional breathlessness as better, the same or worse. | 2 weeks
Quality of life as assessed by SGRQ and the hospital anxiety and depression score | 2 weeks
Sense wear activity monitor measures of daily number of steps walked, daily expenditure and time spent at different levels of activity. | 1 week
Continuous oxygen saturation for 48 hours at weekly intervals | 48 hours
Individual questions specifically related to activity from both the k-BILD and the SOBQ questionnaires | 2 weeks
Qualitative assessment of the impact of ambulatory oxygen | 2 weeks of treatment
  semi-structured open-ended interviews in a subset of 20 patients and their carers

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Renzoni, Dr, Study Chair — RB&HFT
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- [Derived] Visca D, Mori L, Tsipouri V, Fleming S, Firouzi A, Bonini M, Pavitt MJ, Alfieri V, Canu S, Bonifazi M, Boccabella C, De Lauretis A, Stock CJW, Saunders P, Montgomery A, Hogben C, Stockford A, Pittet M, Brown J, Chua F, George PM, Molyneaux PL, Margaritopoulos GA, Kokosi M, Kouranos V, Russell AM, Birring SS, Chetta A, Maher TM, Cullinan P, Hopkinson NS, Banya W, Whitty JA, Adamali H, Spencer LG, Farquhar M, Sestini P, Wells AU, Renzoni EA. Effect of ambulatory oxygen on quality of life for patients with fibrotic lung disease (AmbOx): a prospective, open-label, mixed-method, crossover randomised controlled trial. Lancet Respir Med. 2018 Oct;6(10):759-770. doi: 10.1016/S2213-2600(18)30289-3. Epub 2018 Aug 28. PMID 30170904
- [Derived] Visca D, Tsipouri V, Mori L, Firouzi A, Fleming S, Farquhar M, Leung E, Maher TM, Cullinan P, Hopkinson N, Wells AU, Banya W, Whitty JA, Adamali H, Spencer LG, Sestini P, Renzoni EA. Ambulatory oxygen in fibrotic lung disease (AmbOx): study protocol for a randomised controlled trial. Trials. 2017 Apr 28;18(1):201. doi: 10.1186/s13063-017-1912-9. PMID 28454553